CLINICAL TRIAL: NCT04264884
Title: Daratumumab Subcutaneous Pre-approval Access Study
Brief Title: Pre-Approval Access for Administration of Daratumumab Subcutaneously (SC) in Participants Who Are Unable to Receive Intravenous (IV) Daratumumab
Status: Approved for marketing | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108780; 54767414MMY4031 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

MeSH Terms: interventions — daratumumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Daratumumab — Daratumumab 1800 milligram (mg) will be administered as a fixed dose by subcutaneous (SC) injection.

SUMMARY:
The purpose of this pre-approval access (PAA) program is to provide treatment to participants with serious/life-threatening diseases or conditions.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC